CLINICAL TRIAL: NCT00141856
Title: Health E Heart Study (South Texas Veterans Health Care System Heart Failure Disease Management Program/Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Bauer, Richard - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 045-0023-313; Bauer0004
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2008-06-23 (Estimated); Status verified 2008-06

CONDITIONS: Heart Failure, Congestive
Keywords: Dis Management; Heart Decompensation; Hearts; Veteran (M01.930)
MeSH Terms: conditions — Heart Failure

ARMS (1):
- 1 (Other)
  Interventions: Behavioral: Telephone care

INTERVENTIONS:
Behavioral: Telephone care

SUMMARY:
The primary objective of this telephonic heart failure specific patient education study is to assess the incremental clinical, psycho-social, and functional lifestyle benefits of the Health E Heart Study (South Texas Veterans Health Care System Heart Failure Disease Management Program/Study) when added to standard care among veteran beneficiaries with a heart failure diagnosis. A secondary objective is to assess the impact of the Health E Heart Study on total system utilization costs.

DETAILED DESCRIPTION:
CHF is one of the most common diagnoses for Department of Veterans Affairs (VA) patients. Cost of care, particularly inpatient hospitalization, is high dollar expenditure in the budget.

Study subjects, recruited from the enrolled patient population of the STVHCS, are identified by a diagnosis of CHF in VA clinical databases. Administrative and clinical inclusion and exclusion criteria will be applied by review of medical records. Subjects who appear to meet inclusion criteria will be mailed a pre-enrollment letter containing an Information Sheet describing the program. A follow-up phone call by an RN will go over the program in detail, review the Information Sheet, and initiate enrollment if the subject wishes to participate. As a less than minimal risk study, verbal consent or refusal will be documented in the respective subject's computerized medical record. Assenting subjects will be randomized by the last digit of the social security (odd and even) in a 1:1 ratio to the control group (standard care at STVHCS) or the intervention group (receiving the telephonic disease management services in addition to standard care). The intervention group will receive a telephonic intervention for one year that consists of formal scheduled nurse telephone education sessions, 24-hour access to a nurse counseling and symptom advice telephone line, printed action plans, workbooks, and individualized assessment letters, medication compliance reminders, vaccination reminders, and physician alerts about signs and symptoms of decompensation. Once enrolled, the RN conducts a telephonic assessment at intake, 6, and 12 months to assess each participant's knowledge, behavior, and health status related to the HF condition.

All subjects enrolled in the study will continue to receive comprehensive heart failure care from the STVHCS with those subjects randomized to the program receiving the additional telephonic intervention. Risk stratification is determined from a combination of review of the medical record patient admission history, and other self-reported information. Factors considered include: Goldman Specific Activity Scale, self-management practices, medical history, medical management, and psychosocial factors. The algorithm employs Boolean logic and sorts patients into one of three categories that determines the frequency of scheduled calls over the course of the year. The communications to physicians occurs through the VA CPRS system regularly, usually after each scheduled patient call. Pre-specific clinical, process, and economic outcomes will be collected on all subjects and analyzed at 6 and 12 months post-randomization.

Comparisons: The study will compare resources consumed in providing care to patients with heart failure post-randomization receiving standard care with resources consumed with standard care supplemented by the Health E Heart Disease Management Program. The study will measure direct VA medical care costs.

Study subjects will all receive comprehensive medical care for congestive heart failure from the STVHCS. Experimental subjects will receive additional telephone calls, patient education sessions, customized treatment and self-management plans, and written patient education materials. All subjects will receive telephonic assessments of health status, and functional status at 6 and 12 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria are designed to enroll a population of VA patients with moderate-severe heart failure who are expected to be reasonably representative of and generalizable to potential candidates for the Health E Heart Disease Management Program intervention. To be eligible for the study, veteran beneficiaries must:

* Be 18 years of age
* Have a diagnosis of heart failure
* Have received care in urgent care or have been hospitalized, or have more than 12 outpatient visits in the last twelve months.
* Speak either English or Spanish.

Exclusion Criteria:

Exclusion criteria are designed to exclude persons who are unable to participate in the intervention, whose mortality or health care utilization are driven by co-morbid conditions, or who are enrolled in other research.

* End-stage renal disease on chronic dialysis
* Prior heart transplant
* End-stage or terminal illness in addition to heart failure, such as metastatic malignancy or AIDS with anticipated life expectancy less than 6 months.
* Residence in a nursing home
* Currently participating in another research or care management program.
* No access to a telephone
* Severe dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2005-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Cardiovascular death/re-hospitalization within 6 to12 months from enrollment; 6 to 12 month all-cause mortality/re-hospitalization treatment failure; 6-month heart failure mortality/re-hospitalization; interim analyses | At 6 months and at 12 months

SECONDARY OUTCOMES:
all measures at 6-month intervals
Secondary outcomes include alternative definitions of clinical impact through chart review at study start; functional status and resource utilization and costs at study start, at 6 months, and at twelve months.

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Bauer, MD MSc BA, Principal Investigator — VA South Texas Health Care System
Locations (1):
- VA South Texas Health Care System, San Antonio, Texas, United States

REFERENCES:
- [Result] Goff DC Jr, Pandey DK, Chan FA, Ortiz C, Nichaman MZ. Congestive heart failure in the United States: is there more than meets the I(CD code)? The Corpus Christi Heart Project. Arch Intern Med. 2000 Jan 24;160(2):197-202. doi: 10.1001/archinte.160.2.197. PMID 10647758
- [Result] Berg GD, Wadhwa S, Johnson AE. A matched-cohort study of health services utilization and financial outcomes for a heart failure disease-management program in elderly patients. J Am Geriatr Soc. 2004 Oct;52(10):1655-61. doi: 10.1111/j.1532-5415.2004.52457.x. PMID 15450041
- [Result] Galbreath AD, Krasuski RA, Smith B, Stajduhar KC, Kwan MD, Ellis R, Freeman GL. Long-term healthcare and cost outcomes of disease management in a large, randomized, community-based population with heart failure. Circulation. 2004 Dec 7;110(23):3518-26. doi: 10.1161/01.CIR.0000148957.62328.89. Epub 2004 Nov 7. PMID 15531765
- [Result] Fonarow GC. Heart failure disease management programs: not a class effect. Circulation. 2004 Dec 7;110(23):3506-8. doi: 10.1161/01.CIR.0000151101.17629.20. No abstract available. PMID 15583088
- [Result] Mendez GF, Cowie MR. The epidemiological features of heart failure in developing countries: a review of the literature. Int J Cardiol. 2001 Sep-Oct;80(2-3):213-9. doi: 10.1016/s0167-5273(01)00497-1. PMID 11578717
- [Result] McCullough PA, Philbin EF, Spertus JA, Kaatz S, Sandberg KR, Weaver WD; Resource Utilization Among Congestive Heart Failure (REACH) Study. Confirmation of a heart failure epidemic: findings from the Resource Utilization Among Congestive Heart Failure (REACH) study. J Am Coll Cardiol. 2002 Jan 2;39(1):60-9. doi: 10.1016/s0735-1097(01)01700-4. PMID 11755288